CLINICAL TRIAL: NCT04599530
Title: A Comprehensive Evaluation of a New Generation Bionic Foot
Brief Title: A Comprehensive Evaluation of a the Talaris Demonstrator
Acronym: TD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jo Ghillebert, Doctorandus, Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VUB-Axiles
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Amputation

STUDY DESIGN:
Intervention Model Description: A within Subject Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Biomechanical (Other): All experimental tasks will be evaluated on biomechanical outcome measures
  Interventions: Device: Talaris Demonstrator
- Psychological (Other): All experimental tasks will be evaluated on psychological outcome measures
  Interventions: Device: Talaris Demonstrator
- Physiological (Other): All experimental tasks will be evaluated on biomechanical outcome measures
  Interventions: Device: Talaris Demonstrator
- Performance (Other): All experimental tasks will be evaluated on biomechanical outcome measures
  Interventions: Device: Talaris Demonstrator

INTERVENTIONS:
Device: Talaris Demonstrator — The Talaris Demonstrator will be evaluated during daily activities and compared to the current prosthesis

SUMMARY:
The Talaris Demonstrator is developed in continuation of previous prototypes called the AMPfoot 2.0, 3.0 and 4.0. The main goal of the experiment is to evaluate the effectiveness of TD during daily activities.

DETAILED DESCRIPTION:
A within study design will be conducted in order to evaluate four different prosthetic devices (current, non-propulsive TDF, propulsive TDF and Cyberlegs) with ten participants.

Prior to the baseline test, a familiarization trial aimed to accustom participants to the experimental protocol, to get used to the measurements and interface of the measurement devices. The baseline experimental trial is implemented to evaluate the current prosthesis during the different tests. The same tests will be performed during the evaluation of the other devices. Participants are asked to perform the following consecutive tasks with ten minutes of rest in between each task. The first task is a stair climbing test where participants' will be asked to ascend and descend a staircase. Participants start in front of the staircase and are asked to ascend and descend as fast as possible. Bilateral handrails are required to allow support when needed. The ascending phase is initiated with the prosthetic side, while the first step of the descending phase is performed with the non-involved leg. The second task is the L-test, where participants are asked to rise from a chair, walk through an office door, turn 90 degrees, walk down a hallway, turn 180 degrees and then return in the same way to the seated position. A total distance of 20 meter will be covered. The slope walking test assesses the participants' ability to ascend and descend an inclined ramp as fast as possible. For safety reasons bilateral handrails are warranted. Participants start the test in an upright position in front of the ramp and are asked to ascend the ramp, turn around on the platform, descend the ramp and return to the starting position. During a two-minute walk test, participants are asked to respond as fast as possible to a stimulus visualized on a computer screen one meter in front of the treadmill. Finally, a hallway six-minute walk test will be performed on a hallway at a self-selected walking speed, which closely relates to the most efficient walking speed.

In between each test with a novel device, participants need accustom to the novel device to ensure a good alignment and fitting. Participants will be fitted and aligned to the novel device by a physiotherapist and prosthetist.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 - 75 years
* Gender: men and women
* Level of amputation: unilateral transfemoral
* Vascular, traumatic, congenital or other cause of amputation
* Completed the rehabilitation program, meaning that participants possess their final prosthesis
* Medicare Functional Classification Level: K2-4
* Participants wear their prosthesis for at least 8 hours/day

Exclusion Criteria:

* Any neurological disease
* No upper limb or bilateral amputation
* Stump pain or bad fit of the socket

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomechanical: step length | 1 year
  Step Length in cm
Biomechanical: cadence | 1 year
  Cadence steps/min
Biomechanical: step width | 1 year
  Step width in cm
Biomechanical: swing phases | 1 year
  in % of gait cycle
Biomechanical: stance phases | 1 year
  in % of gait cycle
Physiological: oxygen consumption | 1 year
  in ml/min/kg
Psychological: Visual Analogue Scale | 1 year
  For Fatigue and Comfort on a scale from 0 to 10
Performance: walking speed | 1 year
  In meter per second
Performance: duration | 1 year
  secondfs

IPD SHARING:
Plan to Share IPD: No